CLINICAL TRIAL: NCT02887469
Title: Efficacy and Safety of Rapid Intermittent Correction Compared With Slow Continuous Correction With Hypertonic Saline in Patient With Moderately Severe or Severe Symptomatic Severe Hyponatremia (SALSA Trial)
Brief Title: Efficacy and Safety of Rapid Intermittent Compared With Slow Continuous Correction in Severe Hyponatremia Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: National Research Foundation of Korea (Other)
Responsible Party: Principal Investigator, Seon Ha Baek, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B1605346003
Record Dates: First submitted 2016-08-01; First posted 2016-09-02 (Estimated); Last update posted 2020-04-09 (Actual); Status verified 2020-04

CONDITIONS: Hyponatremia Symptomatic
Keywords: Hyponatremia; Hypertonic saline; Treatment; Osmotic demyelination syndrome
MeSH Terms: conditions — Hyponatremia | interventions — Saline Solution, Hypertonic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intermittent bolus group (Active Comparator): <<Within 6hr>>
  * Moderately Severe : 3% saline 2ml/kg over 20min *1 (unknown bwt 100ml)
  * Severe :3% saline 2ml/kg over 20min *2 (unknown bwt 100ml)
  <additional treatment> Repeat 3% saline 2ml/kg over 20min at every sample time point (at 1/6hr) till Na 5-9 mmol/L inc from initial Na and sx relief
  <<During 6-24hr>>
  - Moderately Severe or Severe
  : Repeat 3% saline 2ml/kg over 20min at every sample time point(at 12/18/24hr) till Na 5-9 mmol/L inc from initial Na and sx relief
  <<During 24-48hr>>
  * Moderately Severe or Severe : Repeat 3% saline 2ml/kg over 20min at every sample time point (at 30/36/42/48hr) till Na 10-17 mmol/L inc from initial Na or Na ≥ 130mmol and sx relief
  Interventions: Drug: 3% hypertonic saline
- slow continuous infusion group (Active Comparator): <<Within 24hr>>
  - Moderately Severe: 3% saline 0.5ml/kg/hr (unknown bwt 25ml/hr)
  - Severe: 3% saline 1ml/kg/hr (unknown bwt 50ml/hr)
  Infusion protocol modification as below by Na at every sample time point (at 1/6/12/18/24 hr)
  If Na 5-9 mmol/L inc from initial Na and sx relief : stop 3% saline infusion regardless of △ Na
  if △ Na inc <0.5mmol/hr or △ Na inc <3mmol/6hr : add 0.25ml/kg/hr, restart 0.5ml/kg/hr if previously stopped
  if △ Na inc ≥0.5mmol/hr or △ Na inc ≥ 3mmol/6hr
  : maintain infusion rate
  <<During 24-48hr>>
  - Moderately Severe and Severe
  Infusion protocol modification as below by Na at every sample time point (at 30/36/42/48hr)
  If Na 10-17 mmol/L inc from initial Na or Na ≥ 130mmol and sx relief
  : stop 3% saline infusion regardless of △ Na
  if △ Na inc <1.5mmol/6hr
  : add 0.25ml/kg/hr or restart 0.25ml/kg/hr if previously stopped
  if △ Na inc ≥ 1.5mmol/6hr
  : maintain infusion rate
  Interventions: Drug: 3% hypertonic saline

INTERVENTIONS:
Drug: 3% hypertonic saline — The same as above

SUMMARY:
This study will investigate efficacy and safety of rapid intermittent correction compared with slow continuous correction with hypertonic saline in patient with moderately severe or severe symptomatic severe hyponatremia

DETAILED DESCRIPTION:
Moderate to severe symptomatic hyponatremia requires prompt treatment with hypertonic saline. The extent and rate of increase in serum sodium (sNa) levels during treatment are critical. Several methods for continuous infusion of hypertonic saline were used to guide rate of fluid administered to achieve the required serum sodium target. As based on static model, they had a bias to over-correction of hyponatremia. Alternative approach to treatment with hypertonic fluid is to use small, fixed boluses to achieve controlled increments in sNa. However, there was no high quality evidence on whether hypertonic saline are best given in continuous infusion (preferred by most) or bolus injection. The aim of present study, a multi-center (Seoul National University Bundang Hospital [2016.8~], Seoul National University Boramae Medical Center [2016. 9~], Hallym University Dongtan Sacred Heart Hospital [2017.7~]), randomized, open labelled, controlled clinical trial, is to investigate efficacy and safety of rapid intermittent correction compared with slow continuous correction with hypertonic saline in patient with moderately severe or severe symptomatic severe hyponatremia. A total 178 patients, who suffer from symptomatic severe hyponatremia, will be enrolled and randomly assigned to receive either intermittent bolus infusion or slow continuous infusion by 3% hypertonic saline. Subjects will take different rate of 3% hypertonic saline for 24-48 hours stratified by severity of clinical symptoms. Serum sodium will be measured at every six hours during two days.

ELIGIBILITY:
Inclusion Criteria:

* In emergency setting (2016.6-) and/or inpatients at ward (2018.9-)
* Glucose corrected serum sodium ≤125 mmol/L
* Patients with moderately severe or severe symptom

  * Moderately severe

    :Nausea without vomiting Drowsy, Headache General weakness, myalgia
  * Severe :Vomiting, Stupor, Seizures, Coma (Glasgow Coma Scale ≤8)
* written consent

Exclusion Criteria:

* Pseudohyponatremia: serum osmolality > 275 mOsm/kg

  - If the serum osmolality is > 275 mOsm/kg but the BUN is ≥ 30 mg/dL, the patients can be registered if calculated serum osmolality (2 x plasma [Na] + [Glucose]/18) is <275 mOsm/kg
* Primary polydipsia: urine osmolality ≤ 100 mOsm/kg
* Glucose corrected serum sodium >125 mmol/L
* Arterial hypotension (SBP <90mmHg and MAP <70mmHg)
* Anuria or urinary outlet obstruction
* Liver disease

  * transaminase levels >3 times the upper limit normal
  * Known LC with ascites or diuretics use or PSE Hx or Varix Hx
* Uncontrolled diabetes mellitus (HbA1C > 9%)
* Women who are pregnant or breast feeding
* History of cardiac surgery excluding PCA, acute myocardial infarction, sustained ventricular tachycardia, ventricular fibrillation, acute coronary syndrome, cebrovascular trauma, and increased intracranial pressure within the 3 months prior to randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2016-08; Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Incidence of overcorrection rate at any given period | up to 48 hours
  Increase in sNa by >12 mmol/L within 24 hours or Increase in sNa by >18 mmol/L within 48 hours All subjects receive hypertonic saline by intermittent bolus or slow continuous infusion for 48 hours, serum Na will be measured.

SECONDARY OUTCOMES:
Rapid improvement of symptoms | up to 24 hours
  Change of symptoms from baseline to 24 hours after hypertonic fluid treatment
Time from treatment initiation to an increase of serum Na ≥ 5 mmol/L | up to 48 hours
Incidence of target correction rate | up to 48 hours
  Target correction rate is defined by achieved serum Na <10 mmol/L within 24 hours, achieved serum Na <18 mmol/L within 48 hours
Time to serum Na >130 mmol/L | up to 48 hours
  Time from treatment initiation to achieved serum Na> 130mmol/L
Length of hospital stay | up to 8 weeks
Incidence of additional treatment | up to 48 hours
  Additional treatment is performed if symptom is not relieved or undercorrection develops (achieved Na < 5mmol/L with 24 hours or achieved Na <12mmol/L within 48 hours)
Incidence of osmotic demyelinating syndrome confirmed by ICD -10 code or MRI | up to 48 hours
Incidence of relowering treatment | up to 48 hours
  Relowering treatment is performed as below if achieved serum Na is <10 mmol/L within 24 hours, achieved serum Na is <18 mmol/L within 48 hours.
  1. discontinuing ongoing active treatment
  2. start infusion of 10ml/kg of 5% dextrose over 1hr ± desmopressin 2mcg IV
Change of Glasgow coma scale (GCS) ≤8 | up to 48 hours
  Change in GCS of hyponatremia symptoms at pretreatment, 24 hours, and 48 hours after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Seon Ha Baek, PhD, Principal Investigator — Hallym University Dongtan Sacred Hospital
Locations (3):
- South Korea (3):
  - Hallym University Dongtan Sacred Hospital, Hwaseong-si, Gyeonggi-do
  - Seoul National University Bundang Hospital Clinical Trial Center, Seongnam-si, Gyeonggi-do
  - Seoul National University Boramae Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Spasovski G, Vanholder R, Allolio B, Annane D, Ball S, Bichet D, Decaux G, Fenske W, Hoorn EJ, Ichai C, Joannidis M, Soupart A, Zietse R, Haller M, van der Veer S, Van Biesen W, Nagler E; Hyponatraemia Guideline Development Group. Clinical practice guideline on diagnosis and treatment of hyponatraemia. Eur J Endocrinol. 2014 Feb 25;170(3):G1-47. doi: 10.1530/EJE-13-1020. Print 2014 Mar. PMID 24569125
- [Derived] Baek SH, Jo YH, Ahn S, Medina-Liabres K, Oh YK, Lee JB, Kim S. Risk of Overcorrection in Rapid Intermittent Bolus vs Slow Continuous Infusion Therapies of Hypertonic Saline for Patients With Symptomatic Hyponatremia: The SALSA Randomized Clinical Trial. JAMA Intern Med. 2021 Jan 1;181(1):81-92. doi: 10.1001/jamainternmed.2020.5519. PMID 33104189
- [Derived] Lee A, Jo YH, Kim K, Ahn S, Oh YK, Lee H, Shin J, Chin HJ, Na KY, Lee JB, Baek SH, Kim S. Efficacy and safety of rapid intermittent correction compared with slow continuous correction with hypertonic saline in patients with moderately severe or severe symptomatic hyponatremia: study protocol for a randomized controlled trial (SALSA trial). Trials. 2017 Mar 29;18(1):147. doi: 10.1186/s13063-017-1865-z. PMID 28356136